CLINICAL TRIAL: NCT04908813
Title: A Randomized, Double-blinded，Multicenter，Phase II Clinical Study of HLX22 (Recombinant Humanized Anti-HER2 Monoclonal Antibody Injection) in Combination With Trastuzumab and Chemotherapy (XELOX) Versus Placebo in Combination With Trastuzumab and Chemotherapy (XELOX) for Treatment of Locally Advanced or Metastatic Gastric Cancer (GC)
Brief Title: Study of HLX22 in Combanition With Trastuzumab and Chemotherapy Versus Placebo in Combination With Trastuzumab and Chemotherapy for Treatment of Locally Advanced or Metastatic Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX22-GC-201
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HLX22(25mg/kg)+Trastuzumab + Chemotherapy (XELOX) (Experimental): Participants receive 25mg/kg HLX22 IV every 3 weeks (Q3W) plus trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance thereafter) IV Q3W in combination with XELOX chemotherapy
  Interventions: Drug: HLX22; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine
- HLX22(15mg/kg)+Trastuzumab + Chemotherapy (XELOX) (Experimental): Participants receive 15mg/kg HLX22 IV Q3W plus trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance thereafter) IV Q3W in combination with XELOX chemotherapy
  Interventions: Drug: HLX22; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine
- Placebo +Trastuzumab + Chemotherapy (XELOX) (Active Comparator): Participants receive placebo IV Q3W plus trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance thereafter) IV Q3W in combination with XELOX chemotherapy
  Interventions: Drug: Placebo; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: HLX22 — IV Q3W D1
  Arms: HLX22(15mg/kg)+Trastuzumab + Chemotherapy (XELOX); HLX22(25mg/kg)+Trastuzumab + Chemotherapy (XELOX)
Drug: Placebo — IV Q3W D1
  Arms: Placebo +Trastuzumab + Chemotherapy (XELOX)
Drug: Trastuzumab — IV Q3W D1
Drug: Oxaliplatin — IV Q3W D1
Drug: Capecitabine — PO Q3W D1-D14

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of HLX22 in the HER2+ Locally Adanved or Metastatic Gastric Cancer as the first-line therapy.This study consists of three periods, screening period (28 days), treatment period and follow-up period (including safety follow-up, survival follow-up).Subjects can be enrolled into this study only if they meet inclusion criteria and do not meet exclusion criteria. The enrolled subjects will receive an intravenous infusion of HLX22/placebo and SOC(standard of care: Trastuzumab + XELOX) once every 3 weeks until the loss of clinical benefit, death, intolerable toxicity, withdrawal of informed consent or other reasons as specified in the protocol(whichever occurs earlier).

DETAILED DESCRIPTION:
HLX22(25mg/kg) or HLX22(15mg/kg) or placebo will be administered intravenously [IV] on day 1 of each 3-week cycle. Trastuzumab (8 mg/kg loading dose, 6 mg/kg maintenance dose) will be administered IV on day 1 of each 3-week cycle. SOC chemotherapy is XELOX (1000 mg/m^2 capecitabine administered orally twice daily [BID] on days 1-14 of each 3-week cycle and 130 mg/m^2 oxaliplatin administered IV on Day 1 of each 3-week cycle).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of previously untreated, locally advanced unresectable or metastatic HER2 positive gastric adenocarcinoma.
* HER2-positive defined as either immunohistochemistry (IHC) 3+ or IHC 2+ in combination with in-situ hybridization positive (ISH+) or fluorescent in-situ hybridization (FISH), as assessed by central review on primary or metastatic tumor
* Has measurable disease as defined by RECIST 1.1 as determined by the IRRC
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Has a life expectancy of greater than 6 months
* Has adequate organ function

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has history of HER2 targeted therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 7 months after the last dose of trial treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per RECIST 1.1 assessed by IRRC(Independent Radiology Review Committee) | Up to 5 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by IRRC or death due to any cause, whichever occurs first. PFS will be determined for each treatment arm
Objective Response Rate (ORR) per RECIST 1.1 assessed by IRRC | Up to 5 years
  ORR is defined as the percentage of participants who have a Complete Response ([CR], disappearance of all evidence of disease) or Partial Response ([PR], regression of measurable disease and no new sites) per RECIST 1.1 as assessed by IRRC. ORR will be determined for each treatment arm.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
  OS is defined as the time from randomization to death due to any cause. OS will be determined for each treatment arm.
Duration of Response (DOR) per RECIST 1.1 assessed by IRRC | Up to 5 years
  For participants who demonstrate CR or PR, DOR is defined as the time from first response (CR or PR) to subsequent disease progression or death from any cause, whichever occurs first. DOR will be determined for each treatment arm
Adverse Events (AE) | Up to 5 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experience an AE will be reported for each treatment arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

REFERENCES:
- [Derived] Li N, Qiu M, Zhang Y, Yang M, Lu L, Li W, Ma Y, Hou X, Sun G, Cai M, Wang J, Lu J, Zhong D, Huo Z, Zhang J, Yin X, Deng J, Liu Z, Pan H, Chen Y, Yang F, Yu H, Li J, Wang Q, Zhu J, Li J. A randomized phase 2 study of HLX22 plus trastuzumab biosimilar HLX02 and XELOX as first-line therapy for HER2-positive advanced gastric cancer. Med. 2024 Oct 11;5(10):1255-1265.e2. doi: 10.1016/j.medj.2024.06.004. Epub 2024 Jul 9. PMID 38986608